CLINICAL TRIAL: NCT02620995
Title: Evaluation of Systemic and Penile Microvascular Endothelial Function and Arterial Pressure After Chronic Administration of Sildenafil in Hypertensive Men With Erectile Dysfunction
Brief Title: Effects of Sildenafil on Penile Vascular Function in Hypertensive Men With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior researcher, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 17663813.4.0000.5272
Record Dates: First submitted 2015-12-01; First posted 2015-12-03 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Arterial Hypertension; Erectile Dysfunction
Keywords: hypertension; endothelial dysfunction; erectile dysfunction; sildenafil
MeSH Terms: conditions — Hypertension; Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypertensive patients (Experimental): Hypertensive patients will receive a single oral dose of sildenafil citrate (100 mg) - acute protocol - and a chronic 30-day treatment with sildenafil citrate (50 mg twice daily) - chronic protocol. Penile and systemic microvascular function will be evaluated before and one hour after acute sildenafil administration and in the end of each treatment period.
  Interventions: Drug: sildenafil citrate
- comparator group (Sham Comparator): Normotensive individuals age-matched to the hypertensive patients will receive only a single dose of sildenafil citrate (100 mg) - acute protocol. Penile and systemic microvascular function will be evaluated before and one hour after sildenafil administration.
  Interventions: Other: comparator group

INTERVENTIONS:
Drug: sildenafil citrate — the hypertensive patients with erectile dysfunction will be treated with sildenafil citrate (100 mg daily) or placebo (crossover design)
  Other Names: Viagra
  Arms: hypertensive patients
Other: comparator group — Normotensive individuals age-matched to the hypertensive patients will receive only a single dose of sildenafil citrate (100 mg) - acute protocol. Penile and systemic microvascular function will be evaluated before and one hour after sildenafil administration.
  Arms: comparator group

SUMMARY:
The study will evaluate the effects of a chronic 30-day treatment with sildenafil citrate on penile and systemic microvascular function as well as in blood pressure.

A control group of normotensive age-matched healthy subjects will serve as a comparator group for normal penile and systemic microvascular function.

DETAILED DESCRIPTION:
Vasculogenic erectile dysfunction (ED) is a highly prevalent health problem that is directly related with increased cardiovascular risk. In this context, phosphodiesterase type 5 inhibitors (PDE5 inhibitors) are indicated in the treatment of ED because these drugs increase bioavailability of the endothelial-dependent potent vasodilator nitric oxide. Thus, these drugs could also induce a reduction in arterial pressure and improve microvascular endothelial function in hypertensive patients.

The primary aim of the study is to investigate the acute and chronic effects of sildenafil citrate (®Viagra) on penile and systemic microvascular function of hypertensive patients presenting with ED. The secondary aim is to evaluate the effects of the treatment on arterial pressure.

The study design is a prospective 2 x 2 cross-over, randomized, double blind clinical trial that will include 75 sexually active hypertensive men (age between 50-70 years) under anti-hypertensive treatment (arterial pressure < 160/100 mmHg) presenting with ED. Erectile function will be evaluated using the International Index of Erectile Function (IIEF-5) questionnaire. Patients with non-vasculogenic ED or diabetes will be excluded from the study. Forty-five age-matched healthy subjects will be included as a comparator group.

The evaluation of systemic microvascular function will be performed in the skin of the forearm and penile microvascular function in the skin of the base of the penis using the non-invasive methodology of laser speckle flowmetry coupled to cutaneous iontophoresis of a vasodilator (acetylcholine).

In the acute protocol, microvascular evaluation will be carried out before and one hour after the oral administration of 100 mg of sildenafil citrate. In the chronic protocol, only hypertensive men will be randomized to receive either or placebo sildenafil 50 mg twice daily for 30 days. After a 30-day washout period the patients will receive the complementary treatment.

The evaluation of penile and systemic microvascular function, as well as ambulatory blood pressure monitoring, will be performed before randomization and in the end of each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* arterial hypertension stage I or II
* erectile dysfunction (vasculogenic)

Exclusion Criteria:

* diabetes
* kidney, liver, neurologic and psychiatric diseases

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Penile microvascular vasodilatory capacity | at the end of a 30-day treatment

SECONDARY OUTCOMES:
Blood pressure levels evaluated using ambulatory blood pressure monitoring | at the end of a 30-day treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo V Tibirica, MD, PhD, Principal Investigator — National Institute of Cardiology - Ministry of Health -Brazil
Locations (1):
- National Institute of Cardiology, Ministry of Health, Brazil, Rio de Janeiro, Brazil